CLINICAL TRIAL: NCT01095588
Title: A Phase I, Single-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel-Arm Study of the Effects of Avanafil on the Pharmacokinetics and Pharmacodynamics of Warfarin in Healthy Male Subjects
Brief Title: Study the Effect of Avanafil on the Pharmacodynamics and Pharmacokinetics of Warfarin in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wesley Day, VP Clinical, Vivus, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TA-016
Record Dates: First submitted 2009-01-06; First posted 2010-03-30 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Erectile Dysfunction
Keywords: ED
MeSH Terms: conditions — Erectile Dysfunction | interventions — avanafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Avanafil (Experimental)
  Interventions: Drug: 200 mg Avanafil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 200 mg Avanafil — 2 X 100mg tablets avanafil
  Arms: Avanafil
Drug: Placebo — 2 tablets
  Arms: Placebo

SUMMARY:
This study is designed to look into the effect of avanafil on blood levels of warfarin and to investigate its effect on prothrombin time/international normalized ratio (INR) in healthy men.

DETAILED DESCRIPTION:
The trial is a single-centre, double-blind, randomized, placebo-controlled, 2-way crossover drug interaction study with at least a 21-day washout period.

Each subject will participate in two sessions in which they will be randomized to receive either 200 mg of avanafil or matching placebo for 9 days. On Day 3 of each period, subjects will receive a single dose of warfarin (25 mg). Following the warfarin dose, pharmacokinetic and pharmacodynamic sampling will be taken over a period of 7 days. Subjects will be discharged on Day 10 following the end-of-period evaluation. There will be a washout of at least 21 days between the warfarin doses. The study medications will be administered with 240 mL of water following an overnight fast of at least 10 hours.

Blood samples (3 mL) for the assessment of R- and S-warfarin concentrations in plasma will be drawn on Day 3 prior to warfarin administration and 0.5, 1, 1.5, 2, 4, 6, 9, 12, 24, 48, 72, 96, 120, 144, and 168 hours after the warfarin administration.

Blood samples (3 mL) for the assessment of avanafil and/or metabolite concentrations will be drawn on Day 3 prior to avanafil (or placebo) administration and at 0.5, 1, and 2 hours post-dose.

Blood samples (4.5 mL) for the assessment of prothrombin time (PT) and international normalized ratio (INR) will be drawn at screening, check-in, on Day 3 prior to warfarin administration and at 6, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours post-dose.

Blood samples (4.5 mL) for collagen-induced platelet aggregation will be drawn on Day 3 prior to warfarin administration and at 1, 4, 6, 12, and 24 hours post-dose.

A blood sample (8.5 mL) for VKORC1 and CYP2C9 genotyping will be drawn at the check-in for Period 1.

The overall blood volume required for this study (assuming direct venipuncture for each sample) will be approximately 446 mL.

All subjects will be confined at the Clinical Research Unit starting in on Day -2 for diet equilibration and will remain confined for approximately 24 hours following the last study drug administration on Day 9.

Adverse events, laboratory evaluations, electrocardiogram, physical examination, and vital signs will be assessed at various times during the study.

ELIGIBILITY:
Inclusion Criteria:

* adult male subjects,
* 21 to 45 years of age,
* must be medically healthy with no clinically significant screening results.

Exclusion Criteria:

* history or clinical evidence of clinically relevant cardiovascular (including thromboembolic disorders), hepatic, renal, hematological, endocrine, pulmonary, gastrointestinal, psychiatric or neurological impairment;
* any clinically significant laboratory abnormalities as judged by the investigator;
* systolic blood pressure < 90 or >120 mmHg;
* diastolic blood pressure < 50 or > 90 mmHg;
* allergy to or previous adverse events with PDE5 inhibitors, warfarin or their constituents;
* use of prescription or over-the-counter drugs that are known to interfere with metabolism by the cytochrome P450 3A4 enzyme within 30 days of screening;
* use of any investigational drug within 30 days of screening; use of any prescription or over-the-counter drugs or herbal remedies within 14 days of screening;
* history of alcohol or drug abuse within 18 months, history of smoking within 6 months;
* positive urine alcohol and drug test;
* positive serum cotinine test;
* positive serology for HIV, HCV, HBsAg.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - PK parameters AUC, C-max and t-max of R-and S-warfarin | 24 hrs
Pharmacodynamics - Prothrombin time, INR values, and area under effect-time curve (AUEC) of prothrombin and INR on days 14 and 15 | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Shiyin Yee, PhD, Study Director — VIVUS LLC